CLINICAL TRIAL: NCT01427777
Title: The Thirty-six-Month Immunogenicity Evaluation of Quadrivalent HPV (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) Vaccine in Chinese Female Subjects Aged 9 to 45 Years and Male Subjects Aged 9 to 15 Years
Brief Title: 3-year Immunogenicity Evaluation of Quadrivalent HPV Vaccine in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangxi Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Rongcheng Li, Director of Vaccine Research Center, Guangxi Center for Disease Control and Prevention
Other Study IDs: V501-030-1
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-09

CONDITIONS: Anogenital Human Papilloma Virus Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HPV Vaccine: People that receive HPV vaccine in V501-030

SUMMARY:
The thirty-six-month immunogenicity evaluation of Quadrivalent HPV (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) Vaccine in Chinese female subjects aged 9 to 45 years and male subjects aged 9 to 15 years.

DETAILED DESCRIPTION:
All eligible subjects will be enrolled for one visit. A medical history and physical examination will be conducted on all subjects. A 10 mL blood specimen will be collected. All Sera should be shipped to PPD Vaccines and Biologics Laboratory in the US. The serum specimen will be tested at PPD Laboratory with competitive Luminex immunoassay (cLIA) and multiplexed HPV immunoassay. The purpose of the quadrivalent HPV cLIA and multiplex is to detect neutralizing antibody and total IgG to HPV virus-like particles (VLPs), serotypes 6, 11, 16, 18, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese subject who participated in V501-030 in Per-protocol population.
* Subject agrees to provide study personnel with a primary telephone number as well as an alternate telephone number for follow-up purposes.
* Subject is willing to give consent/assent.

Exclusion Criteria:

* Subject is concurrently enrolled in clinical studies of investigational agents which may interfere with the evaluation of the study objectives.
* Subject has any condition which in the opinion of the investigator might interfere with the evaluation of the study objectives
* Subject has a history of known prior vaccination with a HPV vaccine, either active agent or placebo after receiving the vaccination during V501-030

Ages: 9 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects who participated in V501-030 in Per-protocol population
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-09; Study Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rongcheng Li, MD, Principal Investigator — Guangxi CDC
Locations (1):
- Liuzhou CDC, Liuchow, Guangxi, China

REFERENCES:
- [Derived] Huang T, Liu Y, Li Y, Liao Y, Shou Q, Zheng M, Liao X, Li R. Evaluation on the persistence of anti-HPV immune responses to the quadrivalent HPV vaccine in Chinese females and males: Up to 3.5 years of follow-up. Vaccine. 2018 Mar 7;36(11):1368-1374. doi: 10.1016/j.vaccine.2018.02.006. Epub 2018 Feb 7. PMID 29428178